CLINICAL TRIAL: NCT05883228
Title: Anesthesiologist Perspectives/Opinions/Ethics on Intraoperative/Intraprocedural Code Status and Intraoperative/Intraprocedural Code Status Management Plans
Acronym: AnesOpIntraDNR
Status: Withdrawn | Type: Observational
Why Stopped: Pre-empted by another survey
Sponsor: Joseph Hendrix (Other)
Responsible Party: Sponsor-Investigator, Joseph Hendrix, Associate Professor of Anesthesiology and Pain Management, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: STU-2023-0329; STU-2023-0329 (Other: UTSW IRB certification approval as EXEMPT)
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Physician's Role; Opinions
Keywords: DNR (Do Not Resuscitate); DNAR (Do Not Attempt Resuscitation); Intraoperative; Intraprocedural; Ethics; Anesthesiologist; Resuscitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This survey aims to understand anesthesiologists' opinions on intraoperative/intraprocedural code status management (like for example, Do Not Resuscitate (DNR)) in various patient scenarios. Your valuable input will help us better understand current practices and preferences in the field.

The understanding of the perspectives of ASA (American Society of Anesthesiologists) member staff anesthesiologists and staff anesthesiologists in general on this matter is of critical importance in the field of anesthesiology as the intraoperative/intraprocedural patient population continues to collectively get older and sicker in the future.

Goal/Aims: The goal of this survey is to ascertain the perspectives of all active ASA member staff anesthesiologists and staff anesthesiologists in general on the matters of intraoperative/intraprocedural code status and intraoperative/intraprocedural code status management plans

DETAILED DESCRIPTION:
Title: Anesthesiologist Perspectives on Intraoperative/Intraprocedural Code Status and Intraoperative/Intraprocedural Code Status Management Plans Introduction: This survey aims to understand anesthesiologists' opinions on intraoperative/intraprocedural code status management in various patient scenarios. Your valuable input will help us better understand current practices and preferences in the field.

Goal/Aims: The goal of this survey is to ascertain the perspectives of all active ASA members on the matters of intraoperative/intraprocedural code status and intraoperative/intraprocedural code status management plans.

Sample Size/Scope: All Active ASA member staff anesthesiologists and staff anesthesiologists in general in the United States of America

Face/Construct Validity:

Are the components of the measure (e.g., questions) relevant to what's being measured? Yes, the questions and structure of the questions are relevant for the intended purpose of ascertaining the respondent's perspectives on intraoperative/intraprocedural code status and intraoperative/intraprocedural code status management plans.

Does the measurement method seem useful for measuring the variable? Yes, the questions and structure of the questions are useful for the intended purpose of ascertaining the respondent's perspectives on intraoperative/intraprocedural code status and intraoperative/intraprocedural code status management plans.

Is the measure seemingly appropriate for capturing the variable? Yes, the questions and structure of the questions are appropriate for capturing the intended purpose of ascertaining the respondent's perspectives on intraoperative/intraprocedural code status and intraoperative/intraprocedural code status management plans.

All questions and question structures are consistent and thematically similar to previous studies/research cited.

Kerry Tanner, Chapter 6 - Survey designs, Editor(s): Kirsty Williamson, Graeme Johanson, Research Methods (Second Edition), Chandos Publishing, 2018, Pages 159-192, ISBN 9780081022207, https://doi.org/10.1016/B978-0-08-102220-7.00006-6.

Geyer ED, Miller R, Kim SS, Tobias JD, Nafiu OO, Tumin D. Quality and Impact of Survey Research Among Anesthesiologists: A Systematic Review. Adv Med Educ Pract. 2020 Aug 25;11:587-599. doi: 10.2147/AMEP.S259908. PMID: 32904509; PMCID: PMC7456338.

Sousa VEC, Dunn Lopez K. Towards Usable E-Health. A Systematic Review of Usability Questionnaires. Appl Clin Inform. 2017 May 10;8(2):470-490. doi: 10.4338/ACI-2016-10-R-0170. PMID: 28487932; PMCID: PMC6241759.

Kash BA, Cheon O, Halzack NM, Miller TR. Measuring Team Effectiveness in the Health Care Setting: An Inventory of Survey Tools. Health Serv Insights. 2018 Aug 24;11:1178632918796230. doi: 10.1177/1178632918796230. PMID: 30158825; PMCID: PMC6109848.

Patient Safety/Quality of Care: The results of this survey will be utilized to inform and empower the greater understanding and implementation of practices regarding intraoperative/intraprocedural code status and intraoperative/intraprocedural code status management plans for future policy matters in the field of anesthesiology.

Priority: The understanding of the perspectives of ASA member staff anesthesiologists and staff anesthesiologists in general on this matter is of critical importance in the field of anesthesiology as the intraoperative/intraprocedural patient population continues to collectively get older and sicker in the future.

ELIGIBILITY:
Inclusion Criteria:

* Active Member of ASA
* Anesthesiologist
* Clinical Practice in United States of America

Exclusion Criteria:

* Participant refusal
* Inability to access survey instrument

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: ASA Active Member Anesthesiologists in the United States of America
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Aggregate Responses to Questions on Survey of ASA Members and Anesthesiologists | One year
  Aggregate Responses to Questions on Survey of ASA Members and Anesthesiologists

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hendrix, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is an anonymous survey study where no individual identifying information is ever captured, stored, or analyzed at any time during the study. Only the aggregate data is captured, stored, and analyzed.

REFERENCES:
- [Background] Clemency MV, Thompson NJ. "Do not resuscitate" (DNR) orders and the anesthesiologist: a survey. Anesth Analg. 1993 Feb;76(2):394-401. PMID 8424522
- [Background] Gu X, Eshkevari L, Powell T, Titus AJ, O'Guin C. Certified Registered Nurse Anesthetists' Management of the Perioperative Do-Not-Resuscitate Order: Evaluating Trends in Required Reconsideration. AANA J. 2021 Dec;89(6):491-499. PMID 34809754
- [Background] Burkle CM, Swetz KM, Armstrong MH, Keegan MT. Patient and doctor attitudes and beliefs concerning perioperative do not resuscitate orders: anesthesiologists' growing compliance with patient autonomy and self determination guidelines. BMC Anesthesiol. 2013 Jan 15;13:2. doi: 10.1186/1471-2253-13-2. PMID 23320623
- [Background] Hiestand D, Beaman M. Perioperative Do-Not-Resuscitate Suspension: The Patient's Perspective. AORN J. 2019 Mar;109(3):326-334. doi: 10.1002/aorn.12612. PMID 30811574
- [Background] Baumann M, Killebrew S, Zimnicki K, Balint K. Do-Not-Resuscitate Orders in the Perioperative Environment: A Multidisciplinary Quality Improvement Project. AORN J. 2017 Jul;106(1):20-30. doi: 10.1016/j.aorn.2017.05.002. PMID 28662781
- [Background] Kim C, Keneally R. The Do Not Resuscitate (DNR) order in the perioperative setting: practical considerations. Curr Opin Anaesthesiol. 2021 Apr 1;34(2):141-144. doi: 10.1097/ACO.0000000000000974. PMID 33630773
- [Background] Baldor DJ, Smyrnios NA, Faris K, Guilarte-Walker Y, Celik U, Torres U. A Controlled Study in CPR-Survival in Propensity Score Matched Full-Code and Do-Not-Resuscitate ICU Patients. J Intensive Care Med. 2022 Oct;37(10):1363-1369. doi: 10.1177/08850666221114052. Epub 2022 Jul 11. PMID 35815880